CLINICAL TRIAL: NCT06374420
Title: Small Airway Disease And Bronchial Hyperreactivity In Patients With Post Acute Covid-19 Syndrome
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Tamer Awad, MD, Mansoura University
Other Study IDs: MD.21.11.564
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this work is to estimate the frequency of small airway disease and/or the bronchial hyperreactivity in follow up of postacute covid survivors.

DETAILED DESCRIPTION:
This is a observational longitudinal study investigating pulmonary sequelae of covid-19.

Study site:

Mansoura university hospital, chest department and post covid outpatient clinic.

Elmahalla chest hospital and outpatients clinic.

Time of study :

Two years from September 2021 to September 2023

Target population:

Adults with confirmed covid 19 who remaining symptomatic after 30 days from the diagnosis.

Sample size The study will include 100 selected cases during period from 2021 to 2023

Patients :

The enrolled patients are adults who survived acute covid-19 and presented for clinical follow up.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory adult patients confirmed diagnosis of covid -19 either on typical CT chest basis or PCR and passed period of acute illness (28 days from start of symptoms) but still with clinical symptoms.

Exclusion Criteria:

* Hospitalized or requiring intensive care unit. Known patients with chronic lung diseases Uncontrolled comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with confirmed covid 19 who remaining symptomatic after 30 days from the diagnosis.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
investigating pulmonary sequelae of covid-19. | 3moth
  The selected post covid patients on the day of their clinic visit (one to three months after being diagnosed covid 19
investigating pulmonary sequelae of covid-19. | 6 month
  The selected post covid patients on the day of their clinic visit (6 months after being diagnosed covid 19

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakhlia, Egypt